CLINICAL TRIAL: NCT04760275
Title: A Sequential Multiple Assignment Randomized Trial (SMART) Assessing Medication and CBT Sequencing Strategies in the Treatment of Predominantly Ethnic Minority, Underserved Youth With Anxiety Disorders
Brief Title: Fluoxetine vs CBT in Childhood Anxiety Disorders
Acronym: SMART
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Bradley Peterson, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-19-00478; 16008 (Other: The Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Fluoxetine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication - Fluoxetine (Active Comparator): Approved medication by the U.S. Food and Drug Administration (FDA) for treating anxiety disorders in children.
  The study's starting dose, and minimum permitted, will be 10 mg/day; should that not be tolerated, the patient will be withdrawn from active treatment (but not from study follow-up). After 1 week at 10 mg/day, the dose will increase to 20 mg/day. After completion of week 4, 10 mg/day dose increases will be permitted every other week as tolerated, up to a maximum daily dose of 80 mg/day. If patients are on doses >20mg/day, the total daily dose can be prescribed either once daily or split into twice daily administrations.
  Interventions: Drug: Fluoxetine
- Cognitive Behavioral Therapy (CBT) (Active Comparator): Type of talk therapy that aims to identify and replace negative thoughts, using positive behavioral skills to create and maintain positive moods and healthy relationships.
  The Coping Cat (CC) program will be used as the behavioral intervention for this study.CC is an established evidence-based CBT treatment for pediatric anxiety. It is delivered in individual therapy sessions with anxious children.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Fluoxetine — This will be a single-blind SMART design of 24 weeks duration that will employ two sequential levels of randomization, one in each of two 12-week stages of the study.
  In Stage 1, participants will be randomized 1:1 to receive 12 weeks of the medication fluoxetine in upward-titrated dosages. In Stage 2, also 12 weeks in duration, participants who remit during the first 12 weeks of treatment will continue maintenance-level therapy with fluoxetine. All participants who do not remit will be randomized (1:1) to either (1) optimization of fluoxetine (increasing the dose of fluoxetine as tolerated), or (2) optimization of fluoxetine and addition of Cognitive Behavioral Therapy (CBT).
  Arms: Medication - Fluoxetine
Behavioral: Cognitive Behavioral Therapy (CBT) — This will be a single-blind SMART design of 24 weeks duration that will employ two sequential levels of randomization, one in each of two 12-week stages of the study.
  In Stage 1, participants will be randomized 1:1 to receive 12 weeks of weekly CBT implemented with Coping Cat (CC). In Stage 2, also 12 weeks in duration, participants who remit during the first 12 weeks of treatment will continue maintenance-level therapy with CBT. All participants who do not remit will be randomized (1:1) to either (1) optimization of CBT (intensifying exposure practice and skills review), or (2) optimization of CBT and addition of the medication fluoxetine.
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
Treatment of every child with anxiety disorder begins with the question of which treatment to start first. Both fluoxetine and CBT have strong empirical support, but few studies have compared their initial effectiveness head-to-head, and none has investigated what to do if the treatment tried first isn't working well-whether to optimize the treatment already begun or to add the other treatment.

Aims of the study:

1. The study will assess whether beginning with Cognitive Behavioral Therapy (CBT) or fluoxetine medication is more effective in improving youth-rated anxiety symptoms over the 24-week intervention
2. If the initial intervention fails to induce clinical remission by week 12, the study will assess whether optimizing the initial treatment modality alone, or adding the other modality to the first, yields better symptom improvement by week 24
3. The study will assess whether one sequence of treatment modalities - i.e., CBT followed by optimized CBT; CBT followed by optimized CBT+ medication; medication followed by optimized medication; medication followed by optimized medication + CBT -- is significantly better or worse than predicted from the two main effects
4. The study will assess the stability of treatment response for ≥12 months following completion of the 24-week trial

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 8-17
* Patients screening positive (score ≥3) on the SCARED-5 (possible range 0-10, higher scores indicate greater severity) and positive (score ≥25) on the SCARED-41 (possible range 0-82, higher scores indicate greater severity).
* Patients with an anxiety disorder (generalized anxiety, separation anxiety, panic, or social anxiety) on the Schedule for Affective Disorders and Schizophrenia for School-Aged Children, computerized version (KSADS-COMP).
* Patients with a score of >8 on the Child Anxiety Impact Scale (CAIS- possible range of scores is 0-81, higher scores indicate greater impact) representing at least moderately severe illness.
* Patients and at least one parent/caregiver of all ages, who are fluent in either English or Spanish.
* Patient and their parent agree for the child to be randomized to either fluoxetine or CBT.

Exclusion Criteria:

* Patients with a neurological disorder or unstable medical condition, as determined by medical chart and medical history review by the site director and PI.
* Females who are pregnant or sexually active but not using an effective method of birth control (potential adverse fetal effects of medication).
* Patients with any of the following characteristics/conditions on the Columbia-Suicide Severity Rating Scale (CSSRS- possible range of scores 0-5, higher scores representing greater severity):

  1. Patients scoring a 3 AND access to crisis level support is unavailable OR
  2. Patients scoring a 4 if frequency, duration, and deterrent all = 1 AND treatment in a specialty mental health clinic is not available OR
  3. Patients scoring a 4 if frequency, duration, OR deterrents are > 1
  4. Patients scoring a 5 4. Due to the cognitive and socio-emotional demands of the CBT protocol, we will exclude youths who are likely to be functioning at a developmental level outside the minimum age for the treatment manual (age 8): Youths who are placed outside of a general education (GE) classroom for > 50% of the school day or require a one-on-one classroom aide to maintain placement in a GE class, or are performing academically below the 2nd grade level in reading and language arts.
* Patients with a current obsessive-compulsive disorder (OCD) diagnosis, for which this study's treatments would be inappropriate clinically and ethically, on the KSADS-COMP.
* Patients with a current post-traumatic stress disorder (PTSD) diagnosis, for which this study's treatments would be inappropriate clinically and ethically, with the following characteristics/conditions on the Child Trauma Screen (CTS) and KSADS-COMP:

  a. Patients scoring at least 1 past trauma on the events portion of the CTS AND a reaction score ≥10 (possible range of scores 0-18, with higher scores representing more severe reactions) on the parent report.
* Patients currently receiving fluoxetine. Those who are currently receiving any other selective serotonin reuptake inhibitor (SSRI), serotonin-norepinephrine reuptake inhibitor (SNRI), other antidepressant, or benzodiazepine for the treatment of either anxiety or sleep disturbance and who otherwise meet all eligibility requirement will be permitted to taper and discontinue their medication to enter the study if they wish to do so and if they otherwise still meet all eligibility requirements after the taper.

Psychopharmacologists on the study team will provide guidelines for the medication taper and discontinuation, but the patient's previously prescribing clinician must first agree that the taper is clinically reasonable and agree to conduct the taper after first discussing the risks and benefits of the taper and discontinuation with the child and parent(s). The study term will not conduct or oversee the medication taper.

* Patients who have taken Monoamine Oxidase Inhibitors (MAOIs), Pimozide, Thioridazine, Olanzapine, Tricyclic Antidepressants (TCAs), Antipsychotics such as Haloperidol and Clozapine, Anticonvulsants such as Phenytoin and Carbamazepine within 2 weeks prior to starting the study.
* Patients currently in foster care.
* Patients currently receiving psychotherapy.

  a. Patients who are receiving psychotherapy and who, together with their parents and treating clinician, agree that it is reasonable either to pause or discontinue their psychotherapy for the duration of the 24-week trial, will be permitted to do so and may then enroll in our SMART study.
* Patients with a past diagnosis of Bipolar Disorder, as determined by medical chart and medical history review by the site director and PI OR Patients who score ≥18 on the Parent General Behavior Inventory-10-Item Mania Scale (PGBI-10M) (possible range 0-30, higher scores representing an increased likelihood of diagnosis).
* Patients with a current/active psychotic diagnosis (schizophrenia, schizoaffective, schizophreniform, psychosis not otherwise specified (NOS), or depression with psychotic features), as determined by medical chart and medical history review by the site director and PI.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Youth - SCARED (Screen for Child Anxiety Related Disorders) | Week 24
  Patient ratings of anxiety symptom severity. Possible range of scores is 0-82, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Parent - SCARED (Screen for Child Anxiety Related Disorders) | Week 24
  Parent ratings of anxiety symptom severity. Possible range of scores is 0-82, with higher scores indicating greater severity.
Youth - Child Anxiety Impact Scale (CAIS) | Week 24
  Patient ratings of anxiety functional impairment. Possible range of scores is 0-81, with higher scores indicating greater impact.
Parent - Child Anxiety Impact Scale (CAIS) | Week 24
  Parent ratings of anxiety functional impairment. Possible range of scores is 0-81, with higher scores indicating greater impact.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S. Peterson, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that are primary and secondary trial outcomes used for the Patient-Centered Outcomes Research Institute (PCORI) Final Research Report.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: When PCORI makes the Final Research Report available on the PCORI website, or at the time of publication of the research project's primary results in a peer-reviewed journal, whichever comes first, and ending 7 years after.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee directed by a PCORI-designated repository. To achieve the stated research purpose underlying the data request approved by the repository. Once a request is approved by an independent review committee, the data requestor's institution must enter into a Data Use Agreement (DUA) with the PCORI-designated repository. The PCORI-designated repository will make the Full Data Package (or required data elements, as applicable) available for third-party requests.
URL: https://www.pcori.org/sites/default/files/PCORI-Policy-for-Data-Management-and-Data-Sharing.pdf

REFERENCES:
- [Derived] Peterson BS, West AE, Weisz JR, Mack WJ, Kipke MD, Findling RL, Mittman BS, Bansal R, Piantadosi S, Takata G, Koebnick C, Ashen C, Snowdy C, Poulsen M, Arora BK, Allem CM, Perez M, Marcy SN, Hudson BO, Chan SH, Weersing R. A Sequential Multiple Assignment Randomized Trial (SMART) study of medication and CBT sequencing in the treatment of pediatric anxiety disorders. BMC Psychiatry. 2021 Jun 30;21(1):323. doi: 10.1186/s12888-021-03314-y. PMID 34193105